CLINICAL TRIAL: NCT01054495
Title: Evaluating Placebo Interventions in Acupuncture Research
Brief Title: Placebo in Acupuncture
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Centre of Complementary and Alternative Medicine, Norway (Other)
Collaborators: Norwegian Acupuncture College (Unknown)
Responsible Party: Arne Johan Norheim, MD PhD, National Research Centre of Complementary and Alternative Medicine, Norway
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2009/1-7
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Nausea; Vomiting
Keywords: Acupuncture; Sham acupuncture; Laser; Methodology; Control intervention; Pilot; Nausea and vomiting in early pregnancy; Patient's experience of different acu-stimulation; Blinding in acupuncture research
MeSH Terms: conditions — Nausea; Vomiting | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture (Active Comparator): Needle acupuncture at acupuncture point pericardium 6
  Interventions: Drug: Acupuncture
- Sham acupuncture (Sham Comparator): Non-penetrating sham needling at acupuncture point pericardium 6
  Interventions: Device: Sham acupuncture
- Laser acupuncture (Placebo Comparator): Laser stimulation at acupuncture point pericardium 6
  Interventions: Device: Laser acupuncture

INTERVENTIONS:
Drug: Acupuncture — The acupuncture needles are inserted in PC 6 bilaterally at the acupuncture point Pericardium 6 (PC6) on each forearm (fig 2). According to the "cun" measurement system of Traditional Chinese Medicine (TCM), the points are located on the palmar surface of anterior forearm at a distance equivalent to the combined width of the women's middle three fingers, proximal to the most prominent wrist crease, and between the tendons of palmaris longus and flexor carpi radialis. We try to keep the depth of the needling to approximately 1,5 cm. At insertion of the acupuncture needle, DeQi is obtained and the needle is then left without any further manipulation/ stimulation (even method) in situ for 15 minutes.
  Arms: Acupuncture
Device: Sham acupuncture — A sham acupuncture needle is placed at PC 6 bilaterally and the tactile stimuli of the skin during the procedure should be obtained. The sham acupuncture needle is then left at site for 15 minutes without any further manipulation/stimulation.
  Arms: Sham acupuncture
Device: Laser acupuncture — A laser is placed in a stand, pointing at PC 6 bilaterally, and left at site for 15 minutes without any further manipulation/stimulation.
  Arms: Laser acupuncture

SUMMARY:
Placebo control in acupuncture research is challenging and difficult. The primary objective of the study is to explore a study design comparing stimulation by real acupuncture needle, sham acupuncture needle and laser. The research question is whether a patient is capable of discriminate different stimulation modality when studying acupuncture stimulation for nausea in early pregnancy. The study is planned as a pilot study including 20 women in each of the three study groups, all-together 60 pregnant women. Intervention will consist of standardised 15 minutes stimulation of acupuncture point pericardium 6 by, either two acupuncture needles, two sham acupuncture needle or two laser devices. All participating women are told that they will get different stimulation at an acupuncture point with potential effect on nausea. The women will record their daily symptoms during a 4 day run-in period, a 3 day intervention period, and thereafter a 4 day follow-up period after treatment in accordance with previous research methodology. In addition, the women will record how they experience the three different stimulations of acupuncture points. The results from the study could be important for planning of future studies where the blinding issue with regard to acupuncture is challenged.

DETAILED DESCRIPTION:
STUDY DESIGN

The study will be a randomized, prospective pilot study testing if acupuncture, sham acupuncture, and laser stimulation all are useful means in preventing nausea and/or vomiting in early pregnancy.

The acu-stimulation will be performed during at a standardised regimen using acupuncture point PC 6 bilaterally. The placebo needle will be placed in the same position at PC 6 bilaterally, however not penetrating the surface of the skin. The third group of women will have a laser pointing at PC 6. All the patients will achieve exactly the same, standardised information and counselling.

Study participants

According to birth rate-statistics there should be approximately 7000 annual pregnancies in Oslo area. Prevalence is estimated to be approximately 0,75. According to this, there should be at least 5000 pregnant women suffering from nausea and/or vomiting each year, and at least 400 each month.

It is likely to assume that only 50 % of pregnant women suffering from nausea and/or vomiting do want any kind of therapy for their complaints (i.e. 200/month). If another 10% of these again respond to advertisements and agree to inclusion in an acupuncture study, this will ensure an adequate number of subjects for the study within the three-month study period.

Recruitment plan

Pregnant women in their first trimester will be recruited through advertisements in media and/or flyers made available by all general practitioners, all pharmacies and all clinics caring for pregnant women.

Randomisation is performed in blocks, in order to eliminate confounders of personnel- or structural nature. In the study we will use a randomisation system with variable block sizes. The randomisation procedure will be preformed by closed envelopes in a row.

TREATMENT PLAN

We wish to administer the anti-nausea therapy at a standardised intervention. The patients will receive all together three sessions on three consecutive days for all three stimulation modalities.

Acupuncture may be associated with adverse effects, but is, nevertheless, regarded as relatively safe when performed according to best practice. However, minor punctuate haemorrhages as well as local discomfort may occur. Any adverse event or side effect is monitored according to registration by the patient.

The women are informed about the study both in a written letter and verbally at time of inclusion. Information is given regarding the use of randomisation and the study focusing on the different stimulation modalities.

60 women are included, divided into three groups:

1. ACUPUNTURE GROUP The acupuncture needles are inserted in PC 6 bilaterally at the acupuncture point Pericardium 6 (PC6) on each forearm (fig 2). According to the "cun" measurement system of Traditional Chinese Medicine (TCM), the points are located on the palmar surface of anterior forearm at a distance equivalent to the combined width of the women's middle three fingers, proximal to the most prominent wrist crease, and between the tendons of palmaris longus and flexor carpi radialis. We try to keep the depth of the needling to approximately 1,5 cm. At insertion of the acupuncture needle, DeQi is obtained and the needle is then left without any further manipulation/ stimulation (even method) in situ for 15 minutes.
2. SHAM ACUPUNCTURE GROUP A sham acupuncture needle is placed at PC 6 bilaterally and the tactile stimuli of the skin during the procedure should be obtained. The sham acupuncture needle is then left at site for 15 minutes without any further manipulation/stimulation.
3. LASER ACUPUNCTURE A laser is placed in a stand, pointing at PC 6 bilaterally, and left at site for 15 minutes without any further manipulation/stimulation.

Effect on nausea and/or vomiting is supposed to occur within minutes or few hours. All women included in the study should record their symptoms in a run-in period of 4 days before therapy (day 1-4). The days of therapy is supposed to be day 5-7. They thereafter record symptoms on the 4 consecutive days (day 8-11).

At enrollment, the women will be asked about background variables as well as factors that possibly could affect the outcome of the research. During the whole study period of 11 days, the women are told to record their symptoms according to previous research methodology.

Participants are asked to make three recordings of their symptoms every evening. The first registration is to determine what problems had had the particular day; 1= no problems, 2=nausea and 3=vomiting, regardless of how often and how many times they vomited. In the second registration, the women are asked to estimate how many hours they had suffered each day. In the third registration the women also estimate an overall evaluation of severity their symptoms on a visual analogue scale (VAS).

Every woman participates in the study for 12 consecutive days consisting of a 4 day run-in period, a 3 day treatment period, a 4 day follow up period, and one last day of an ending interview.

The programme for these days is:

Day 0: Day of contact. The woman starts registration of symptoms the next day. Day 1-4: The women register their symptoms every evening. Day 5: Randomization. Day 5-7: The women are treated once daily with one of the three treatments they are randomized to get. The women register how they experience the stimulation of the acupuncture points within one hour after the treatment. The women also register their symptoms of nausea and vomiting every evening. Day 8-11: The women register their symptoms every evening. Dag 12: The woman is phoned and asked to participate in an ending interview.

Data will also be collected with regard to how the women experienced the three different stimulations of the acupuncture points, how and if they obtained the needle-feeling (De Qi), and how and if the consider the treatment effected their condition. The patients are also asked to state credibility of the stimulation and to describe DeQi.

ELIGIBILITY:
Inclusion Criteria:

* Positive urine test for pregnancy by the patients themselves or by their doctor.
* Gestational length of 7-12 weeks estimated according to the Naegele method.
* Nausea related to pregnancy must have lasted for at least one week

Exclusion Criteria:

* Any pre-pregnant underlying disease predisposing for nausea
* Women who has been pregnant by infertility treatment
* The woman can not be treated in hospital for nausea or other diseases during pregnancy.
* Women with any pregnancy related disease or abnormalities discovered at regular pregnancy follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To determine the importance of best practice of point stimulation with regards to the patient's experience of different acu-stimulation. | imidiately after treatment

SECONDARY OUTCOMES:
To evaluate the effectiveness of different acu-stimulation for nausea and vomiting in early pregnancy. | 4 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arne Johan Norheim, PhD, Principal Investigator — The National research center in Complementary and Alternative Medicine
Locations (2):
- Norway (2):
  - The National Research Center in Complementary and Alternative Medicine, Tromsø, Tromso
  - Norwegian Acupuncture College, Oslo